CLINICAL TRIAL: NCT01242826
Title: A Trial Investigating the Pharmacokinetic Properties of Biphasic Insulin Aspart 50 (BIAsp 50) in Healthy Chinese Subjects
Brief Title: Investigation of the Pharmacokinetic Properties of Biphasic Insulin Aspart 50 in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-3881; U1111-1116-2307 (Other: WHO)
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: biphasic insulin aspart 50

INTERVENTIONS:
Drug: biphasic insulin aspart 50 — A single dose of 0.3 U/kg BIAsp 50 for subcutaneous (under the skin) injection

SUMMARY:
This trial is conducted in Asia. The aim of this clinical trial is to investigate the pharmacokinetic properties (the rate at which the trial drug is eliminated from the body) after a single subcutaneous (under the skin) injection of biphasic insulin aspart 50 (BIAsp 50). In addition, the safety and tolerability of BIAsp 50 will be observed

ELIGIBILITY:
Inclusion Criteria:

* Considered generally healthy upon completion of medical history, physical examination, vital signs and electrocardiogram (ECG), as judged by the Investigator (the Physician)
* Body Mass Index (BMI): 19.0-24.0 kg/m2 (both inclusive)

Exclusion Criteria:

* Clinically significant abnormal haematology, biochemistry, lipids or urinalysis screening tests, as judged by the Investigator (the Physician)
* A history of any illness that, in the opinion of the Investigator (the Physician), might confound the results of the trial or a pose risk in administering the trial product to the subject
* Subject who has donated any blood or plasma in the past month or more than 400 mL within 3 months prior to screening (trial entry)
* Not able or willing to refrain from smoking during the inpatient period

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin aspart concentration-time curve from 0 to 24hours | 24 hours profile after single dose of trial drug

SECONDARY OUTCOMES:
Area under the serum insulin aspart concentration-time curve between different time intervals | 24 hours profile after single dose of trial drug
Maximum observed serum insulin aspart concentration | 24 hours profile after single dose of trial drug
Number of adverse events. | After 3-10 days of treatment
Number of hypoglycaemic events | After 3-10 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Beijing, Beijing Municipality, China

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com